CLINICAL TRIAL: NCT03410862
Title: Phase IV Study Evaluating The Safety And Clinical Efficacy Of Elderberry Extract In Patients With Influenza: A Randomized, Double-Blind Placebo-Controlled Trial
Brief Title: Evaluating The Safety And Clinical Efficacy Of Elderberry Extract In Patients With Influenza
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: michael macknin (Other)
Collaborators: Pharmacare Laboratories (Industry)
Responsible Party: Sponsor-Investigator, michael macknin, Staff Physician, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-1682
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Influenza, Human
Keywords: Elderberry; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — elderberry extract; black elderberry extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elderberry Extract (Experimental): Patients will be supplied a liquid Elderberry Extract used to treat their confirmed human influenza. The dosage of the assigned medication will be 15 ml, or 1 tablespoon. Participants aged 5-12 will be asked to take the medication 2 times per day (morning/night) for a period of 5 days. Participants aged 13 and above will be asked to take the medication 4 times per day (morning/noon/afternoon/night) for a period of 5 days.
  Interventions: Drug: Elderberry Extract
- Placebo (Placebo Comparator): Patients will be supplied a liquid Placebo medication (similar in appearance and taste of Elderberry Extract) used to treat their confirmed human influenza. The dosage of the assigned medication will be 15 ml, or 1 tablespoon. Participants aged 5-12 will be asked to take the medication 2 times per day (morning/night) for a period of 5 days. Participants aged 13 and above will be asked to take the medication 4 times per day (morning/noon/afternoon/night) for a period of 5 days.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Elderberry Extract — Thick reddish-brown liquid of Sambucus Nigra (Black Elderberry)
  Other Names: Sambucol
  Arms: Elderberry Extract
Drug: Placebos — Thick reddish-brown liquid similar in appearance and taste to Elderberry Extract not containing elderberry
  Arms: Placebo

SUMMARY:
This research is being done to determine if an extract of cooked elderberries will help decrease the duration and severity of influenza symptoms in patients with confirmed influenza. Involvement in this study requires an initial patient screening at the time of their Emergency Department visit in order to confirm eligibility for the study. Once patients have been consented and enrolled as a participant, they will be randomized to take by mouth either Elderberry Extract or a placebo (a similar appearing and tasting liquid without elderberry) for a duration of 5 days. Study information regarding medication adherence, body temperature, symptoms, severity of symptoms, and any possible side effects will be collected from daily phone surveys conducted by the study coordinator. Participation in the study will end after at least 5 days once the patient has not had a temperature above 100°F and has had no influenza symptoms for at least 24 hours, or after 21 days in the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* With 48 hours or less of an influenza illness documented by polymerase chain reaction
* Have AT LEAST 2 of the following 7 influenza symptoms (nasal congestion, sore throat, cough, aches and pains, fatigue, headaches, and chills or sweats) graded as either moderate or severe
* Have access to a phone
* Subjects are capable of giving informed consent or have an acceptable legally authorized representative capable of giving consent on the subject's behalf with informed assent given by subject.
* Have been prescribed or offered a prescription for oseltamivir (Tamiflu)

Exclusion Criteria:

* Known allergy to elderberry extract or oseltamivir
* Use of antibiotic or antiviral medication on presentation to the study
* Women who are pregnant, breastfeeding women, or do not agree to appropriate contraception (abstinence, hormonal, intrauterine device, and barrier) to prevent pregnancy during the study.
* Patients with HIV
* Patients with cystic fibrosis
* Patients taking elderberry extract

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data, needs HIPPA clearance and specific IRB approval, we did not plan on original data being shared

REFERENCES:
- [Derived] Macknin M, Wolski K, Negrey J, Mace S. Elderberry Extract Outpatient Influenza Treatment for Emergency Room Patients Ages 5 and Above: a Randomized, Double-Blind, Placebo-Controlled Trial. J Gen Intern Med. 2020 Nov;35(11):3271-3277. doi: 10.1007/s11606-020-06170-w. Epub 2020 Sep 14. PMID 32929634

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Elderberry Extract | Placebo
Started | 43 | 44
Completed | 41 | 42
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elderberry Extract | Placebo | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 18 | 34
  Between 18 and 65 years | 27 | 26 | 53
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 38
  Male | 27 | 22 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 16 | 31
  White | 27 | 20 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 8 | 8
Region of Enrollment [Number; unit: participants]
  United States | 43 | 44 | 87

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Until Alleviation of Flu Symptoms Post Treatment
Description: Symptoms will be recorded using the scoring system described in a meta-analysis of "all published and unpublished Roche-sponsored randomized placebo-controlled, double-blind trials of oseltamivir treatment in adult influenza" (BMJ 4/9/2014). "The primary outcome will be time to alleviation of all symptoms. Seven influenza symptoms (nasal congestion, sore throat, cough, aches and pains, fatigue, headaches, and chills or sweats)" will be graded by severity as "none/absent" (0), "mild" (1), "moderate" (2), or "severe" (3). Alleviation will be defined to arise when all symptoms scored as absent or mild, and remain so for at least 21.5 hours."
Time Frame: every 24 hours post study drug administration for minimum of 5 days up to 21 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Elderberry Extract | Placebo
Number analyzed (Participants) | 43 | 44
days | 5.3 (3.6) | 4.9 (2.8)

2. Primary Outcome: Number of Days Until Complete Resolution of All Flu Symptoms for 24 Hours
Description: Participants were called daily and asked to report on the severity of their symptoms present. Symptoms graded according to severity score (NONE/ABSENT=0 MILD=1 MODERATE=2 SEVERE=3).
Time Frame: every 24 hours post study drug administration for minimum of 5 days up to 21 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Elderberry Extract | Placebo
Number analyzed (Participants) | 43 | 44
days | 8.6 (3.9) | 8.7 (3.9)

ADVERSE EVENTS:
Time Frame: Baseline + 6 months
Arm/Group | Elderberry Extract | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/43 | 2/44
Other Adverse Events (participants affected / at risk) | 4/43 | 1/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elderberry Extract (N=43) | Placebo (N=44)
Hospitalization (General disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elderberry Extract (N=43) | Placebo (N=44)
Dry Mouth (General disorders) | 4 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
Outcomes relied solely on self reports of patients' symptoms. We did not subtype the influenza viruses detected in our study and did not check for virus sensitivity to elderberry and to oseltamivir.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT03410862/Prot_SAP_000.pdf